CLINICAL TRIAL: NCT01215331
Title: Gestational Diabetes Mellitus: Insulin or Oral Hypoglycemic Agents?
Brief Title: Gestational Diabetes: Insulin or Oral Hypoglycemic Agents?
Acronym: DG5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Jean-Luc Ardilouze, Endocrinologist, researcher, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-057
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational Diabetes Mellitus; Treatment; Insulin; Metformin; Glyburide
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance | interventions — Insulin; Metformin; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin (Active Comparator): Rapid acting insulin and long acting insulin
  Interventions: Drug: Insulin
- Oral Hypoglycemic Agents (Experimental): Metformin + glyburide + insulin if needed
  Interventions: Drug: Metformin, glyburide and insulin

INTERVENTIONS:
Drug: Insulin — Insulins most commonly used during pregnancy by our group are rapid acting insulins and long acting human insulins (long acting analogs are not authorized in pregnancy). An ultra-fast acting insulin will be started before a meal (1, 2 or 3 meals) at 4-6 IU (according to the weight) if the glycemic value 2 hours after this meal is ≥ 6.7 mmol/L in 50% of cases. It will be increased by 2 units every 2 days until obtaining the aimed objectives. Long acting insulin will be started at 4-6 units at bedtime if the glycemic value before breakfast is ≥ 5.3 mmol/L in 50% of cases, and it will be increased by 2 units every 2 days until reaching the objective. A combination of both insulins could be necessary (maximum of 4 injections per day).
  Arms: Insulin
Drug: Metformin, glyburide and insulin — Metformin (tablets of 500 mg) will be started at 250 mg/day x 1 day, and increased thereafter by 250 mg per day every 3 days until obtaining an adequate glycemic control. If metformin does not prove its effect at a dose of 750 mg, or if the side effects (mainly gastric) command to slow down or not to increase the posology, glyburide will be added.
  Glyburide (tablets of 5 mg) will be started at a dose of 2.5 mg and will be increased by 2.5 mg every 3 days until obtaining an adequate glycemic control. The maximal dose in the study will bw 10 mg. It corresponds to the half of the maximal dose recommended in Canada.
  Treatment failure is defined as glycemia above the Canadian Diabetes Association therapeutic objectives in spite of maximal doses or whether the doses can not be increased because of side effects. Insulin will be added to oral hypoglycemic agents.
  Arms: Oral Hypoglycemic Agents

SUMMARY:
Gestational diabetes mellitus takes place in 2 steps. First, it is the consequence of insulin resistance due to the modifications of the pregnancy hormonal environment, and second, of the deficiency of the beta cells of the pancreas to respond by a sufficient insulin secretion. This physiopathology is closely connected to the one of type 2 diabetes. Insulin, indeed, can remedy these 2 etiologies, but it is logical to think about using oral hypoglycemic agents which have been created to treat them: they are a natural choice because they improve insulin sensitivity (metformin, a biguanide) or insulin secretion (glyburide, a sulfonylurea). It also seems natural to use them in combination, glyburide being added to metformin if needed.

OUR GENERAL RESEARCH HYPOTHESIS IS THAT: in pregnant women with gestational diabetes mellitus, using both oral hypoglycemic agents (glyburide added to metformin if needed) allows a glycemic control comparable to the one obtained with insulin, but with a better acceptability from women and a better health status, diabetes treatment satisfaction and well-being and a reduced postnatal depression.

ELIGIBILITY:
Inclusion Criteria:

* women,
* age ≥ 18 yrs,
* with gestational diabetes at 24-28 weeks (Canadian Diabetes Association (CDA) criteria),
* who need a pharmacological treatment following the failure of the diet and exercise,
* to understand and read French or English.

Exclusion Criteria:

* known type 1 or type 2 diabetes,
* treatment interfering with glucose metabolism,
* allergies to one of the components of the treatment,
* hepatic or hematologic diseases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Glycemic control | 36 and 37th week of gestation
  Mean of the capillary glycemic control at 36 and 37th week of gestation.

SECONDARY OUTCOMES:
Acceptability of the treatment | 8-12 weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Ardilouze, MD, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche clinique du CHUS, Sherbrooke, Quebec, Canada